CLINICAL TRIAL: NCT03058159
Title: Sleep Inertia and Functional Connectivity Between Brain Regions at Awakening : a Functional Magnetic Resonance Imaging (fMRI) Study
Brief Title: Sleep Inertia and Functional Connectivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0675
Record Dates: First submitted 2017-02-09; First posted 2017-02-20 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subjects with a high dream recall frequency (Other)
  Interventions: Other: fMRI
- Subjects with a law dream recall frequency (Other)
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — fMRI scans will be acquired before and after a 40 min nap slot in the afternoon. Functional connectivity between brain region will be assessed analyzing the scans with the CONN toolbox of the Statistical Parametric Mapping (SPM) software.

SUMMARY:
The aim of the study is to investigate the functional connectivity between the brain regions of the default mode network before and after a 40 min nap slot in the afternoon. The hypothesis is that connectivity between brain regions will be decreased after the nap as compared to before the nap.

ELIGIBILITY:
Inclusion Criteria:

* 65 > age > 18
* high or law dream recall frequency

Exclusion Criteria:

* history of psychiatric or neurologic or sleep pathologies
* counter indication for MRI

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Measure: Change of correlation values between the BOLD (Blood Oxygenation Level Dependent) signal time series of the brain regions of the default mode network (DMN) between the scans before and after the nap slot. | fMRI scans will be acquired 5 min before, 5 min after and 25min after the nap slot.
  The hypothesis is that connectivity between the brain regions of the default mode network will be decreased after the nap as compared to before the nap and that it will be more the case for subjects with a high dream recall frequency as compared to subjects with a law dream recall frequency. fMRI scans will be acquired before and after a 40 min nap slot in the afternoon. Functional connectivity between brain region will be assessed analyzing the scans with the functional connectivity toolbox (CONN) of the Statistical Parametric Mapping (SPM) software.

CONTACTS AND LOCATIONS:
Overall Officials: Alain NICOLAS, MD, Principal Investigator — CH le VINATIER
Locations (1):
- CH le VINATIER, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vallat R, Meunier D, Nicolas A, Ruby P. Hard to wake up? The cerebral correlates of sleep inertia assessed using combined behavioral, EEG and fMRI measures. Neuroimage. 2019 Jan 1;184:266-278. doi: 10.1016/j.neuroimage.2018.09.033. Epub 2018 Sep 14. PMID 30223060